CLINICAL TRIAL: NCT05158296
Title: A Double-Masked, Randomized, Controlled, Multiple-Dose Study to Evaluate the Efficacy, Safety and Tolerability of Ultevursen in Subjects With Retinitis Pigmentosa (RP) Due to Mutations in Exon 13 of the USH2A Gene (Sirius)
Brief Title: Study to Evaluate the Efficacy Safety and Tolerability of Ultevursen in Subjects With RP Due to Mutations in Exon 13 of the USH2A Gene (Sirius)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQ-421a-003; 2021-002729-74 (EudraCT Number)
Record Dates: First submitted 2021-11-23; First posted 2021-12-15 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2022-12

CONDITIONS: Retinitis Pigmentosa; Usher Syndrome Type 2; Deaf Blind; Retinal Disease; Eye Diseases; Eye Diseases, Hereditary; Eye Disorders Congenital; Vision Disorders
Keywords: Retinitis Pigmentosa; USH2A; RP; exon 13; RNA therapies; antisense oligonucleotide; exon skipping; Sirius; IVT; mutations in exon 13 of the USH2A gene; NSRP; Non-Syndromic RP; Inherited Retinal Disorders; Usher Syndrome; Intravitreal Injection; ultevursen
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Vision Disorders | interventions — Intravitreal Injections

STUDY DESIGN:
Intervention Model Description: Double-masked, randomized, controlled, multiple-dose study. Subjects will be randomized to one of three treatment groups:
  1. Group 1: Ultevursen 180/60 µg (180 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter)
  2. Group 2: Ultevursen 60/60 µg (60 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter; n = 27)
  3. Group 3: Sham-procedure (administered on Day 1, Month 3 and every 6 months thereafter; n = 27)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subject, site staff (study coordinator, imaging technician, etc) and Investigator will be completely masked. Physician performing IVT and post-IVT monitoring will know if subject is receiving sham or treatment, but will be masked to the dose level. Pharmacist is the only site staff that will be completely unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ultevursen 60/60 µg (Experimental): 60 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter
  Interventions: Drug: Ultevursen
- Ultevursen 180/60 µg (Experimental): 180 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter
  Interventions: Drug: Ultevursen
- Sham-procedure (Sham Comparator): Sham-procedure (no experimental drug administered) on Day 1, Month 3 and every 6 months thereafter
  Interventions: Other: Sham-procedure

INTERVENTIONS:
Drug: Ultevursen — RNA antisense oligonucleotide for intravitreal injection
  Other Names: RNA antisense oligonucleotide for intravitreal injection
  Arms: Ultevursen 180/60 µg; Ultevursen 60/60 µg
Other: Sham-procedure — Sham-procedure (no experimental drug administered)
  Arms: Sham-procedure

SUMMARY:
The purpose of this study is to evaluate the efficacy safety and tolerability of ultevursen administered via intravitreal injection (IVT) in subjects with Retinitis Pigmentosa (RP) due to mutations in exon 13 of the USH2A gene.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy safety and tolerability of ultevursen administered via intravitreal injection (IVT) in subjects with Retinitis Pigmentosa (RP) due to mutations in exon 13 of the USH2A gene.

The below dose levels of ultevursen will be evaluated with the loading dose administered at Day 1 and maintenance dose administered at Month 3 and every 6 months thereafter:

1. Loading dose of 60 µg, maintenance dose of 60 µg
2. Loading dose of 180 µg, maintenance dose of 60 µg

Dose levels will include subjects randomized to sham-procedure or treatment with ultevursen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age OR a minor (12 to < 18 years) with permission from a parent or legal guardian. The lower age limit for pediatric populations is subject to local regulatory and ethics committee requirements.
2. An adult willing to comply with the protocol, follow study instructions, attend study visits as required and willing and able to complete all study assessments. OR A minor able to complete all study assessments and comply with the protocol and has a parent or caregiver willing and able to follow study instructions, and attend study visits with the subject as required.
3. Clinical presentation consistent with RP with Usher syndrome type 2 or nonsyndromic form of RP (NSRP), based on ophthalmic, audiologic, and vestibular examinations.
4. A molecular diagnosis of homozygosity or compound heterozygosity for 1 or more pathogenic exon 13 mutations in the USH2A gene, based on genetic analysis at screening.
5. BCVA between ≥30 and ≤68 letters (approximate Snellen equivalent 20/250 - 20/50) in the treatment eye using the mean BCVA reading at screening. Subjects with a mean BCVA between >68 and ≤73 letters will be allowed with documented historic evidence of a BCVA equivalent decline of >5 letters in both eyes.
6. BCVA between ≥30 and ≤73 letters (approximate Snellen equivalent 20/250 - 20/40) in the contralateral eye (CE), using the mean BCVA reading at Screening.
7. A difference in mean BCVA readings at Screening between the TE and CE of

   ≤10 letters (based on ETDRS). BCVA differences between eyes that are greater than 10 letters may be allowed however, the Investigator should discuss the case with the Medical Monitor.
8. Stable BCVA in the TE and CE, defined as 2 separate BCVA measurements at Screening that fall within ≤ 5 letters for each respective eye.
9. A visible EZ layer on SD-OCT in the TE, as determined by the Investigator.
10. No limitations to SD-OCT image collection that would prevent high quality, reliable images from being obtained in both eyes, as determined by the Investigator.
11. Reliable BCVA, perimetry, and other measurements in both eyes, as described in the Study Reference Manual and Imaging Manual and determined by the Investigator.
12. No visually significant ocular media opacities and adequate pupillary dilation to permit good quality retinal imaging in both eyes, as assessed by the Investigator.

Exclusion Criteria:

1. Presence of additional non-exon 13 USH2A pathogenic mutation(s) on the USH2A allele carrying the exon 13 mutation in subjects who have monoallelic exon-13 mutations.
2. Presence of non-exon 13 USH2A pathogenic mutation(s) on both USH2A alleles in subjects who have biallelic exon 13 mutations.
3. Presence of pathogenic mutations in genes (other than the USH2A gene) associated with Usher syndrome Type 2 or NSRP, or other inherited retinal degenerative diseases or syndromes. Note: The confirmed presence of homozygous or compound heterozygous known disease-causing mutations in other genes involved in recessive retinal dystrophies (RD), or the confirmed presence of known disease-causing mutations in genes involved in dominant or X-linked retinal dystrophies is exclusionary.
4. Presence of any significant ocular (in either eye) or non-ocular disease/disorder (or medication and/or laboratory test abnormalities) which, in the opinion of the Investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or the subject's ability to participate in the study. This includes but is not limited to a subject who has uncontrolled cystoid macular edema (CME). CME is permissible if stable for 3 months (with or without treatment). Past CME is permissible if resolved for more than 1 month.
5. History or presence of ocular herpetic diseases (including herpes simplex virus, varicella zoster or cytomegalovirus) in either eye.
6. Presence of any active ocular infection in either eye.
7. Presence of any of the following lens opacities in the study eye: cortical opacity ≥

   +2, posterior subcapsular opacity ≥ +2, or a nuclear sclerosis ≥ +2, and which are: 1) clinically significant in the opinion of the Investigator, 2) would adequately prevent clinical and photographic evaluation of the retina.
8. History of amblyopia in either eye that resulted in significant vision loss, in the opinion of the Investigator.
9. Receipt within 3 months prior to Screening of any intraocular or periocular surgery (including refractive surgery), or an IVT injection or planned intraocular surgery or procedure in either eye during the course of the study. For YAG laser treatment of a posterior capsular opacity, receipt within 1 month prior to Screening or planned procedure in either eye during the course of the study.
10. Current treatment or treatment within the past 12 months with therapies known to influence the immune system (including but not limited to steroid implants, cytostatics, interferons, tumor necrosis factor (TNF)-binding proteins, drugs acting on immunophilins, or antibodies with known impact on the immune system). Subjects that have been treated with systemic steroids within the past 12 months or that require intermittent use of topical steroids may be considered for inclusion following approval by the Medical Monitor.
11. A history of glaucoma or an IOP greater than 21 mmHg in either eye that is not controlled with medication or surgery. IOP measurements between 21 and 24 mmHg may be allowed however, the Investigator should discuss the case with the Medical Monitor.
12. Use of any investigational drug or device within 90 days or 5 half-lives preceding the first dose of study medication, whichever is longer, or plans to participate in another study of an investigational drug or device during the course of the study.
13. Any prior treatment with genetic or stem-cell therapy for ocular or non-ocular disease.
14. History of malignancy within 2 years prior to Screening, except adequately treated squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
15. Known hypersensitivity to antisense oligonucleotides or any constituents of the injection.
16. Pregnant and breastfeeding subjects. Females of childbearing potential and males must comply with using highly effective methods of contraception as defined in the protocol. Women of non-childbearing potential may be included without the use of adequate birth control.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepul Bio Medical Monitor, Study Director — Sepul Bio; Sepul Bio Clinical Operations Director, Study Director — Sepul Bio
Locations (15):
- United States (10):
  - Shiley Eye Institute - UC San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore, Maryland
  - Center for Clinical Research Operations, Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin
- Universitaetsklinikum Tuebingen Department für Augenheilkunde, Tübingen, Germany
- Netherlands (2):
  - RadboudUMC, Nijmegen
  - Het Oogziekenhuis Rotterdam, Rotterdam
- United Kingdom (2):
  - Oxford Eye Hospital, Headington, Oxford
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultevursen 60/60 µg | Ultevursen 180/60 µg | Sham-procedure
Started | 2 | 3 | 2
Completed | 0 | 0 | 0
Not Completed | 2 | 3 | 2
Not completed — Sponsor Decision | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultevursen 60/60 µg | Ultevursen 180/60 µg | Sham-procedure | Total
Number analyzed (Participants) | 2 | 3 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 6
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (1.4) | 47.3 (20.5) | 56.0 (4.2) | 51.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 0 | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 2 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Genotype [Count of Participants; unit: Participants] — Presence of homozygous or heterozygous mutations in the USH2a gene.
  Participants
    Homozygous | 0 | 0 | 1 | 1
    Heterozygous | 2 | 3 | 1 | 6
Phenotype [Count of Participants; unit: Participants] — Subjects were stratified based on phenotype presentation of their retinitis pigmentosa (RP). Syndromic RP, known as Usher syndrome type 2, is associated with congenital moderate to severe hearing loss, and later detection of the retinal disease (ie, RP). Non-syndromic RP is not associated with other signs and symptoms as part of a genetic syndrome.
  Participants
    Syndromic | 2 | 2 | 2 | 6
    Non-Syndromic | 0 | 1 | 0 | 1
Baseline Best Corrected Visual Acuity (BCVA) - Treated Eye [Mean (Standard Deviation); unit: letters] — Baseline Best Corrected Visual Acuity (BCVA) is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) vision chart after mandatory manifest refraction.
  letters | 53.0 (14.1) | 54.7 (11.1) | 59.0 (11.3) | 55.4 (10.1)
Baseline Best Corrected Visual Acuity (BCVA) - Contralateral Eye [Mean (Standard Deviation); unit: letters] — Baseline Best Corrected Visual Acuity (BCVA) is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) vision chart after mandatory manifest refraction.
  letters | 61.0 (5.7) | 71.0 (11.3) | 68.5 (2.1) | 67.4 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: Mean change from baseline in best corrected visual acuity(BCVA) based on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart
Time Frame: 18 months of treatment versus sham-procedure
Population: Zero participants were analyzed due to premature study termination, per Sponsor decision for reasons unrelated to safety. No subject enrolled reached the primary endpoint target of 18 months, therefore no data is available for analysis.
Arm/Group | Ultevursen 60/60 µg | Ultevursen 180/60 µg | Sham-procedure
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Proportion of Patients Who Maintain Vision Defined by BCVA Loss Less Than 15 Letters (ETDRS)
Description: Proportion of patients who maintain vision defined by BCVA loss less than 15 Letters based on ETDRS
Time Frame: 27 months
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Other Analyses of Best Corrected Visual Acuity (BCVA)
Description: Change from baseline in other analyses of Best Corrected Visual Acuity (BCVA)
Time Frame: 27 months
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Ellipsoid Zone (EZ) Area and Width as Imaged by Spectral Domain Optical Coherence Tomography (SD-OCT)
Description: Change from baseline in ellipsoid zone (EZ) area and width as imaged by spectral domain optical coherence tomography (SD-OCT)
Time Frame: 27 months
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Low Luminance Visual Acuity (LLVA)
Description: Change from baseline in Low Luminance Visual Acuity (LLVA)
Time Frame: 27 months
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Microperimetry
Description: Change from baseline in Microperimetry
Time Frame: 27 months
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in Full-field Stimulus Threshold (FST)
Description: Change from baseline in Full-field Stimulus Threshold (FST)
Time Frame: 27 months
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in PRO Measures
Description: As assessed by the Veteran Affairs Low Vision Visual Functioning Questionnaire (VA LV VFQ-20), Patient Global Impressions of Severity (PGI-S) and Patient Global Impressions of Change (PGI-C)
Time Frame: 27 months
Reporting Status: Not Posted

9. Secondary Outcome: Ocular and Non-ocular Adverse Events (AEs)
Description: Ocular and non-ocular adverse events (AEs)
Time Frame: 27 months
Reporting Status: Not Posted

10. Secondary Outcome: Cmax of Ultevursen in Serum
Description: Maximum concentration (Cmax) of ultevursen in serum
Time Frame: 27 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 10 months for each participant. Study was terminated prematurely, therefore follow-up maximum range is first patient first visit to last patient last visit.
Description: Any event/condition noted once the subject receives their first dose of study drug until the End of study visit (30 days +/- 14 days post last dose of study drug).
Arm/Group | Ultevursen 60/60 µg | Ultevursen 180/60 µg | Sham-procedure
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 2/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultevursen 60/60 µg (N=2) | Ultevursen 180/60 µg (N=3) | Sham-procedure (N=2)
Conjunctival haemorrhage (Eye disorders) | 1 | 2 | 0
Eye pain (Eye disorders) | 1 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study prematurely terminated due to sponsor decision for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall be free to publish, present, or use any Data and results arising out of its performance of the protocol. At least 30 days prior to submission for publication, institution shall submit to Sponsor for review and comment any proposed oral or written publication. Institution will consider any such comments in good faith but is under no obligation to incorporate Sponsor's suggestions. The review period for abstracts or poster presentations shall be 30 days.

DOCUMENTS (2):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT05158296/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT05158296/SAP_001.pdf